CLINICAL TRIAL: NCT02471391
Title: A Phase 2 Study of ABT-199 in Combination With Ibrutinib in the Treatment of Patients With Relapsed or Refractory Mantle Cell Lymphoma (AIM Study)
Brief Title: ABT-199 & Ibrutinib in Mantle Cell Lymphoma (AIM)
Acronym: AIM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14/148
Record Dates: First submitted 2015-05-12; First posted 2015-06-15 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — venetoclax; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ibrutinib + ABT-199 (Experimental)
  Interventions: Drug: ABT-199; Drug: Ibrutinib

INTERVENTIONS:
Drug: ABT-199
Drug: Ibrutinib

SUMMARY:
This research will test the combination of two new drugs, called ibrutinib and ABT199, taken together in the treatment of Mantle Cell Lymphoma. Other studies have indicated the potential for these drugs to be used in the treatment of participants with Mantle Cell Lymphoma. In this study, the investigators will test the combination of the two drugs together, in order to determine what effects (good and bad) it has on mantle cell lymphoma.

This study has two phases. The first phase is the Primary Evaluation Phase and will closely monitor the effects of ibrutinib and ABT199 for a period of 13 months. Participants who complete 13 months of treatment and continue benefiting from the study treatments will be allowed to continue both drugs until progression or intolerance in the Continuation Phase. The purpose of this phase is to provide patients with continuing access to both ibrutinib and ABT199. Patients will receive routine care from clinician, who will record any sideeffects that may be experienced.

This is one of the first trials in the world to study the combination of ibrutinib and ABT199 together. Therefore the effectiveness of the combination of the study drugs will be assessed, as will how they affect mantle cell lymphoma and how it develops resistance to the treatments. The investigators also do not know whether combining the two drugs together will cause unexpected side effects. Therefore, the study will monitor patients closely and perform scans, blood tests, bone marrow biopsies and other tests at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be >/= 18 years of age.
2. Subject must have a confirmed diagnosis of Mantle Cell Lymphoma (MCL) according to WHO (2008) criteria, and have received at least one prior line of systemic therapy for MCL.
3. Subject requires treatment in the opinion of the investigator, and has at least one site of radiographically assessable disease not previously irradiated (lymph node with largest diameter >/= 1.5cm, or unequivocal hepatomegaly / splenomegaly)
4. Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of </= 2.
5. Subject must have adequate bone marrow function at Screening as follows:

   * Absolute Neutrophil Count (ANC) >/= 1.0 x 109/L (neutropenia due to marrow infiltration may be supported by growth factors);
   * Platelets >/= 50 x 109/L (entry platelet count must be independent of transfusion within 7 days).
6. Subject must have adequate coagulation, renal, and hepatic function, per laboratory reference range at Screening as follows:

   * aPTT and PT not to exceed 1.5 × the upper limit of normal (ULN);
   * Serum creatinine not to exceed 2 x ULN, and a calculated creatinine clearance of at least 50 mL/min using the Cockcroft-Gault equation or a 24-hour urine collection;
   * AST or ALT </= 3.0 × the upper normal limit (ULN) of institution's normal range; Bilirubin </= 1.5 × ULN. Subjects with documented Gilbert's Syndrome may have a bilirubin > 1.5 × ULN.
7. Female subjects of childbearing potential and non-sterile male subjects (with partners of child bearing potential) must practice at least one of the following methods of birth control with partner(s) from initial study drug administration to 90 days after the last dose of study drug:

   * Total abstinence from sexual intercourse as the preferred life style of the subject; periodic abstinence is not acceptable;
   * Surgically sterile partner(s); acceptable sterility surgeries are: vasectomy, bilateral tubal ligation, bilateral oophorectomy or hysterectomy;
   * Intrauterine device (IUD);
   * Double-barrier method (contraceptive sponge, diaphragm or cervical cap with spermicidal jellies or cream AND a condom);
   * Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration.
8. Female subjects of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [B-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study
9. Male subjects must agree to refrain from sperm donation, from initial study drug administration until 90 days after the last dose of study drug.
10. Subject is able to swallow whole tablets.
11. Subject (or their legally-acceptable representatives) must sign an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

Exclusion Criteria:

1. Subject has undergone an allogeneic stem cell transplant within the last 6 months or currently has active graft-vs-host disease requiring the use of immunosuppressants.
2. Subject has active and uncontrolled autoimmune cytopenias (for 2 weeks), including autoimmune hemolytic anemia (AIHA) and immune thrombocytopenic purpura (ITP).
3. Subject has known central nervous system involvement by MCL.
4. Subject previously participated in an ibrutinib clinical trial or subject previously received a Bruton's tyrosine kinase (BTK) inhibitor other than ibrutinib
5. Subject has received the following within 30 days prior to the first dose of study drug:

   •Monoclonal antibody given with anti-neoplastic intent.
6. Subject has received any of the following within 14 days prior to the first dose of study drug, or has not recovered to less than CTC grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapy:

   * Any anti-cancer therapy including chemotherapy, or radiotherapy;
   * Investigational therapy, including targeted small molecule agents.
7. Subject has received the following within 7 days prior to the first dose of study drug:

   •Steroid therapy given with anti-neoplastic intent
8. Subjects requires ongoing therapy with:

   * Potent CYP3A inhibitors (such as indinavir, ketoconazole, and clarithromycin),
   * Potent CYP3A inducers (e.g., rifampin, phenytoin, carbamazepine or St. John's Wort),
   * Warfarin, or or equivalent vitamin K antagonist (eg, phenprocoumon),
   * Antiretroviral medications.
9. Subject has consumed the following within 3 days prior to the first dose of study drug.

   * Grapefruit, or
   * Grapefruit products, or
   * Seville oranges (including marmalade containing Seville oranges), or
   * Star fruit
10. Subject has clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
11. Subject has a life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.

    •specifically, a subject with history of stroke or intracranial hemorrhage within 6 months prior to enrollment is excluded
12. Subject has a history of other active malignancies other than MCL within the past 2 years prior to study entry, with the exception of:

    * Adequately treated in situ carcinoma of the cervix uteri,
    * Adequately treated basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin,
    * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
13. Subject has known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
14. Received live, attenuated vaccines within 4 weeks of first dose of ibrutinib
15. Major surgery within 4 weeks of first dose of ibrutinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Complete response measured using IWG at 16 weeks | Measured at 16 weeks after commencement of treatment.

SECONDARY OUTCOMES:
Completing 4, 16, 28, 40 and 56 weeks of treatment | Assessed at 4, 16, 28, 40 and 56 weeks
Toxicities measured using CTCAE version 4 | Continuously measured while on treatment up to a maximum of 56 weeks
Overall response (CR + PR) using IWG criteria at 4, 16, 28, 40 and 56 weeks | Assessed at 4, 16, 28, 40 and 56 weeks
Complete response using IWG criteria at 4, 16, 28, 40 and 56 weeks | Assessed at 4, 16, 28, 40 and 56 weeks
Minimal residual disease (MRD) at 4, 16, 28, 40 and 56 weeks | Assessed at 4, 16, 28, 40 and 56 weeks
Progression free survival | From start of treatment until the date of first documented progression or date of death from any cause, whichever occures first, assessed up to the date when the last patient has their 13 months assessment.
Overall survival | From start of treatment until the date of death from any cause assessed up to the date when the last patient has their 13 months assessment.
Duration of response | From first disease response date to the date of earliest recurrance or PD, assessed up to the date when the last patient has their 13 months assessment.
Time to progression | From start of treatment until the date of first documented progression assessed up to the date when the last patient has their 13 months assessment.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria

REFERENCES:
- [Derived] Handunnetti SM, Khot A, Blombery P, Burbury K, Thompson PA, Ritchie D, Hicks RJ, Burke G, Koldej RM, Bressel M, Di Iulio JL, Westerman DA, Lade S, Roberts AW, Seymour JF, Tam CS, Anderson MA. Venetoclax and ibrutinib induces durable clinical responses in marginal zone lymphoma. Blood Adv. 2025 Dec 11:bloodadvances.2025016646. doi: 10.1182/bloodadvances.2025016646. Online ahead of print. PMID 41380113
- [Derived] Handunnetti SM, Anderson MA, Burbury K, Thompson PA, Burke G, Bressel M, Di Iulio J, Hicks RJ, Westerman D, Lade S, Pott C, Agarwal R, Koldej R, Ritchie D, Dreyling M, Dawson MA, Dawson SJ, Seymour JF, Roberts AW, Tam CS. Seven-year outcomes of venetoclax-ibrutinib therapy in mantle cell lymphoma: durable responses and treatment-free remissions. Blood. 2024 Aug 22;144(8):867-872. doi: 10.1182/blood.2023023388. PMID 38662991
- [Derived] Davis JE, Handunnetti SM, Ludford-Menting M, Sharpe C, Blombery P, Anderson MA, Roberts AW, Seymour JF, Tam CS, Ritchie DS, Koldej RM. Immune recovery in patients with mantle cell lymphoma receiving long-term ibrutinib and venetoclax combination therapy. Blood Adv. 2020 Oct 13;4(19):4849-4859. doi: 10.1182/bloodadvances.2020002810. PMID 33031542
- [Derived] Tam CS, Anderson MA, Pott C, Agarwal R, Handunnetti S, Hicks RJ, Burbury K, Turner G, Di Iulio J, Bressel M, Westerman D, Lade S, Dreyling M, Dawson SJ, Dawson MA, Seymour JF, Roberts AW. Ibrutinib plus Venetoclax for the Treatment of Mantle-Cell Lymphoma. N Engl J Med. 2018 Mar 29;378(13):1211-1223. doi: 10.1056/NEJMoa1715519. PMID 29590547